CLINICAL TRIAL: NCT01647854
Title: Introduction and Operation of a Mobile Telemedicine System to Support Paramedics in the Emergency Medical Service
Brief Title: Operation of a Mobile Telemedicine System in the EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 005-1003-0034-5; PtJ-Az.: z0909im002b (Other Grant/Funding Number: PTJ)
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Prehospital Emergency; Teleconsultation; Safety
Keywords: emergency medical service; telemedicine; teleconsultation; safety
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: Teleconsultation (Experimental): If patients give informed consent the paramedics can use this system to contact a so called "tele-EMS physician" with an audio-connection to the EMS team who receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. Also 12-lead-ECGs can be transmitted to the tele-EMS physician. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, ECG diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The safety and efficacy of the introduction and operation of this system should be evaluated.
  Interventions: Procedure: Teleconsultation

INTERVENTIONS:
Procedure: Teleconsultation — Teleconsultation in prehospital emergencies

SUMMARY:
The aim of the study is to investigate the safety and efficacy of the operation of a prehospital teleconsultation system in the Emergency Medical Service.

DETAILED DESCRIPTION:
Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. The paramedics can use this system to contact a so called "tele-EMS physician" after consent of the patient is obtained. The tele-EMS physician has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. Also 12-lead-ECGs can be transmitted to the tele-EMS physician. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, ECG diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The safety and efficacy of the introduction and operation of this system should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* prehospital emergency
* consent of the patient for teleconsultation was obtained or patient is unable to consent due to the severity of the emergency

Exclusion Criteria:

* patient refuses consent for teleconsultation
* psychiatric emergency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rate of complications | up to 2 hours
  The incidence of complications due to delegated medications should be evaluated.

SECONDARY OUTCOMES:
Time intervals | up to 2 hours
  on-scene time of EMS, contact (EMS) to hospital arrival time
Duration of teleconsultation | up to 2 hours
  Analysis of the time requirement for teleconsultation with respect to the different EMS districts and different emergencies as well as over time.
Requirement of on-scene EMS physician | up to 2 hours
  Analysis of the requirement of an on-scene EMS physician in respect to the different emergencies and districts.
Technical assessments | up to 2 hours
  Analysis of the technical performance of the system

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital Aachen, Germany, Department of Anesthesiology; Jörg C Brokmann, Dr., Principal Investigator — University Hospital Aachen, Germany, Emergency Department
Locations (1):
- University Hospital Aachen, Aachen, Germany